CLINICAL TRIAL: NCT05427318
Title: Peers Plus Mobile App for Treatment in HIV (PATH)
Brief Title: Peers Plus Mobile App for Treatment in HIV
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01DA053167 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Telemedicine; Substance use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH Active Intervention Arm (Active Comparator): Participants assigned to this group will receive care as usual if they are assigned to this group. In addition, participants in this arm will receive HIV care support from a trained peer navigator and have access to a mHealth web application designed to support their health and HIV care.
  Interventions: Behavioral: PATH
- Usual Care (No Intervention): Participants assigned to this group are in the control arm and will receive standard of care following the Ryan White model of care.

INTERVENTIONS:
Behavioral: PATH — The intervention integrates two theoretically-grounded interventions - one with a strong peer navigator component and the other with a scalable mHealth component - into the intervention called Peers plus mobile App for Treatment in HIV (PATH)
  Other Names: Camino
  Arms: PATH Active Intervention Arm

SUMMARY:
This study called "Peers plus mobile App for Treatment in HIV (PATH)" is a two-arm randomized controlled trial (RCT) evaluating the efficacy of an intervention that combines peer navigation and mobile health (mHealth) technology to support HIV care outcomes among Hispanic and Black Persons Living with HIV (HBPLH).

DETAILED DESCRIPTION:
PATH is a community-academic collaboration with a federally qualified health center serving patients in South San Diego under the Ryan White model of care.

The scientific premise of this RCT is that combining two interventions developed by this team (peer navigation + mHealth) into a single mHealth peer navigation intervention (PATH) will eliminate the need for in-person support from peer navigators, promote high impact on HIV care continuum outcomes, as well as extend broader reach to underserved communities.

The RCT will test the efficacy of PATH with 375 HBPLH (among whom >33% will report stimulant and/or opioid use in the past 6 months).

Aim 1. Improve the primary outcomes - sustained viral suppression (i.e., suppressed viral load at both 6- and 12-month follow-up), and secondary outcomes (e.g., retention in care) compared to usual care.

Sub-aim 1: Explore subgroup differences in efficacy based on factors like race/ethnicity and substance use.

Aim 2. Examine the theory-informed mediators (e.g., self-efficacy to engage in HIV care, HIV stigma) through which PATH has the greatest impact on sustained viral suppression among HBPLH.

Aim 3. Explore whether PATH significantly affects substance-related outcomes (e.g., frequency of substance use, engagement in substance abuse treatment) when compared to usual care among those using substances (i.e., stimulants and/or opioids).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Can read and speak English or Spanish
* Self-reported diagnosis of HIV by a physician or healthcare provider
* Currently prescribed HIV medication
* Having access to an internet browser on a home computer, tablet, or smart phone
* Does not plan to move out of the San Diego area in the next 12 months
* Meets one or more of the following medical chart verified or self-reported criteria

  * One or more detectable viral load test result (>200 copies m/L) in the past 12-months while on antiretroviral therapy for at least 3 months
  * Having missed 1 or more scheduled HIV care appointments in the last 12 months
  * Last HIV care visit was more than 6 months ago
  * Self-reporting less than 90% antiretroviral therapy adherence in the last 4 weeks using the Wilson-3 scale
  * Report stimulant or opioid use (non-prescription) in the past 6 months

Exclusion Criteria:

* <18 years old
* Currently enrolled in any program, intervention, or research study designed to improve antiretroviral therapy adherence or engagement in HIV care (e.g., LinkPositively)
* Members of one of the community advisory boards providing advisement on the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Viral suppression | 6 months
  Having an undetectable HIV viral load; <200 copies/mL
Viral suppression | 12 months
  Having an undetectable HIV viral load; <200 copies/mL

SECONDARY OUTCOMES:
Retention in HIV care | 6 months
  Health Resources and Services Administration definition: ≥ 2 HIV medical visits at least 90 days apart
Retention in HIV care | 12 months
  Health Resources and Services Administration definition: ≥ 2 HIV medical visits at least 90 days apart
Gap in HIV medical visits | 6 months
  Health Resources and Services Administration definition: no HIV medical visits in last 6 months
Gap in HIV medical visits | 12 months
  Health Resources and Services Administration definition: no HIV medical visits in last 6 months
Antiretroviral therapy adherence | 3 months
  Continuous measure of antiretroviral therapy adherence using the Wilson's three-item Adherence Self-Report Scale scale (0-100; 100=perfect adherence)
Antiretroviral therapy adherence | 6 months
  Continuous measure of antiretroviral therapy adherence using the Wilson's three-item Adherence Self-Report Scale scale (0-100; 100=perfect adherence)
Antiretroviral therapy adherence | 9 months
  Continuous measure of antiretroviral therapy adherence using the Wilson's three-item Adherence Self-Report Scale scale (0-100; 100=perfect adherence)
Antiretroviral therapy adherence | 12 months
  Continuous measure of antiretroviral therapy adherence using the Wilson's three-item Adherence Self-Report Scale scale (0-100; 100=perfect adherence)

CONTACTS AND LOCATIONS:
Locations (1):
- San Ysidro Health, San Ysidro, California, United States

REFERENCES:
- [Derived] Pitpitan EV, Horvath KJ, Aldous J, Stockman JK, Patterson TL, Liang M, Barrozo C, Moore V, Penninga K, Smith LR. Peers plus mobile app for treatment in HIV (PATH): protocol for a randomized controlled trial to test a community-based integrated peer support and mHealth intervention to improve viral suppression among Hispanic and Black people living with HIV. Trials. 2024 Mar 22;25(1):212. doi: 10.1186/s13063-024-08042-8. PMID 38520030